CLINICAL TRIAL: NCT03580135
Title: Postoperative Pain Evaluation of Mineral Trioxide Aggregate and Propolis After Pulpotomy in Carious Primary Molars: A Randomized Controlled Trial
Brief Title: Postoperative Pain Evaluation of Mineral Trioxide Aggregate and Propolis After Pulpotomy in Carious Primary Molars
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rawda Nader Mahmoud, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Rawda N.Mahmoud
Record Dates: First submitted 2018-06-09; First posted 2018-07-09 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Pulp Disease, Dental
Keywords: pulpotomy; primary molars; propolis
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Propolis; mineral trioxide aggregate; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Propolis powder (Experimental): * resin (50%),
  * vegetable Balsam, wax
  * essential aromatic oils (30%)
  * salivary secretions (10%)
  * pollen(5%)
  * other substances (5%) including amino acids
    ,ethanol vitamin A, B complex, and E, minerals, steroids
  * ﬂavonoids. The most important pharmacologically active constituents in propolis are ﬂavonoids, which are well-known compounds which have antioxidant, anti-bacterial, antifungal, antiviral, and anti-inﬂammatory properties.
  * Other ingredients: carob powder (free flow agent). Contains no yeast, salt, sugar, starch, milk, preservatives or colors.
  Interventions: Drug: Propolis
- Mineral Tri Oxide (Active Comparator): * Consists of calcium oxide and silicon dioxide.When these raw materials are blended, they produce tricalcium silicate, dicalcium silicate, tricalcium aluminate, and tetracalcium aluminoferrite.
  * A radiopacifier (bismuth oxide) is added to the cement for dental radiological diagnosis.
  Interventions: Drug: Mineral Trioxide Aggregate

INTERVENTIONS:
Drug: Propolis — One and half gram of Standardized Propolis Extract powder (Y.S. Eco Bee Farms Propolis Powder) at 100% was mixed with 1.75 mL of polyethylene glycol (Continental Chemicals, New Delhi, India) to form a thick consistency on a clean dry glass slab with a metal spatula. The paste was carried to the pulp stumps with a metal carrier and then condensed lightly to a thickness of 2 - 3 mm followed by placement of thick mix of GIC to seal the cavity and covered by st.st crown.
  Other Names: propolis bee resin
  Arms: Propolis powder
Drug: Mineral Trioxide Aggregate — MTA paste will be prepared as per the manufacturers' instructions to obtain a putty-like consistency. The mixture will be delivered to the pulp stumps and condensed lightly with a moistened sterile cotton pellet to ensure a thickness of 2 to 3 mm. A thick mix of glass ionomer cement (GIC) will applied over the MTA and covered by st.st crown.
  Other Names: MTA
  Arms: Mineral Tri Oxide

SUMMARY:
The study will be self-funded by investigator and carried out on patients from outpatient clinic in Pediatric Dentistry and Public Health Department- Faculty of Dentistry, Cairo University- Egypt. The procedures will be carried out by postgraduate student Rawda Nader Fathy who has B.D.S. (2011) -Alexandria University- Egypt. The procedures will be carried out on a Knight Midmark Biltmore dental unit (Midmark Corporation 1700 S. Patterson Blvd. Suite 400 Dayton, Ohio 45409, USA) in the post graduate clinic of Pediatric Dentistry and Public Health Department- Faculty of Dentistry, Cairo University- Egypt.

ELIGIBILITY:
Inclusion Criteria:

1. Cooperative patient
2. Healthy 5-8 years old patient with at least one carious primary molar tooth at each side of the patient's mouth.
3. Presence of at least two-thirds of the root length radiographically.
4. Restorable tooth.
5. No signs of hyperemia and hemostasis will be adequately achieved with moistened cotton pellet within 5 minutes after coronal pulp amputation.

Exclusion Criteria:

1. Teeth showing clinical and radiographic evidence of pulp degeneration such as history of spontaneous or nocturnal pain, tenderness to percussion or palpation, pathologic mobility, swelling or fistulous tract, periodontal ligament (PDL) space widening, internal root resorption, external root resorption, furcal radiolucency/inter- radicular bone destruction and/or periapical bone destruction.
2. Patients eliciting history of known allergy to pollens associated with propolis.
3. Parent or guardian refusal to participate.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of postoperative pain after pulpotomy by asking patient and/or parents (binary yes or no) | 9 months
  Binary (yes or no)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data will be available within 9 months completion of study
Access Criteria: data Access will be reviewed by external independent review panel
URL: http://register.clinicaltrials.gov

REFERENCES:
- [Background] Alolofi H, El-Sayed M, Taha S. Clinical and radiographical evaluation of propolis and thymus vulgaris extracts compared with formocresol pulpotomy in human primary molars. BDJ Open. 2016 Jul 29;2:16005. doi: 10.1038/bdjopen.2016.5. eCollection 2016. PMID 29607066
- [Background] Hugar SM, Kukreja P, Hugar SS, Gokhale N, Assudani H. Comparative Evaluation of Clinical and Radiographic Success of Formocresol, Propolis, Turmeric Gel, and Calcium Hydroxide on Pulpotomized Primary Molars: A Preliminary Study. Int J Clin Pediatr Dent. 2017 Jan-Mar;10(1):18-23. doi: 10.5005/jp-journals-10005-1400. Epub 2016 Dec 5. PMID 28377649